CLINICAL TRIAL: NCT01554566
Title: Metabolic Effects of Honey in Type 1 Diabetes Mellitus: a Cross Over Randomised Controlled Pilot Study
Brief Title: Metabolic Effects of Honey in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mamdouh abdulmaksoud abdulrhman, Professor, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: honey1010
Record Dates: First submitted 2012-03-09; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: honey; diabetes; lipids; c-peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Honey; pteropsin, Apis mellifera

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- honey, no honey (Experimental)
  Interventions: Dietary Supplement: honey

INTERVENTIONS:
Dietary Supplement: honey — The subjects in the I/C group consumed 0.5 ml honey/kg/day in the first 12-week period (period 1) while the subjects in the C/I group did not receive honey as a control in period 1. After period 1 the subjects of each group exchanged their protocol for the following 12-week period (period 2).
  Other Names: bee honey

SUMMARY:
This study aimed at evaluation of the metabolic effects of honey, as a supplemental food, in patients suffering from type 1 diabetes mellitus. A crossover design (two 12-weeks intervention periods) was used to measure honey effects. The subjects were randomized into two groups (intervention to control [I/C] and control to intervention [C/I] groups. Each group consisted of 10 patients. . The subjects in the I/C group consumed 0.5 ml honey/kg/day in the first 12-week period (period 1) while the subjects in the C/I group did not receive honey as a control in period 1. After period 1 the subjects of each group exchanged their protocol for the following 12-week period (period 2).

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 1 diabetes mellitus with their last HbA1C less than 10% were candidates for this study.

Exclusion Criteria:

* Coexisting renal or hepatic impairment
* Coexisting diseases e.g., malignancy, other endocrine disorders
* Patients on steroid therapy or other drugs that may affect the body weight or serum lipids.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
serum lipids | 12 wk
  Fasting serum lipids (cholesterol, triglycerides, low density lipoprotein cholesterol and high density lipoprotein cholesterol) were measured at base line, cross over (12 wk) and end point of the study (24 wk)

SECONDARY OUTCOMES:
C-peptide | 12 week
  Fasting and 2 hr postprandial C-peptide were measured at base line, cross over (12 wk) and end point of the study (24 wk)

CONTACTS AND LOCATIONS:
Overall Officials: Mamdouh AM Abdulrhman, professor, Principal Investigator — pediatric department, faculty of medicine, ain shams university; Mohamed H El Hefnawy, professor, Principal Investigator — national institute of diabetes and endocrinology, cairo, egypt; Rasha H Aly, assist. prof, Principal Investigator — pediatric department, faculty of medicine, ain shams university; Rania H Shatla, lecturer, Principal Investigator — pediatric department, faculty of medicine, ain shams university; Doaa M Mohamed, M.B.B.Ch, Principal Investigator — pediatric department, faculty of medicine, ain shams university; Waheed S Mohamed, M.B.B.Ch, Principal Investigator — pediatric department, faculty of medicine, ain shams university
Locations (1):
- National Institute of Diabetes and Endocrinology, Cairo, Kasr El Ainy, Egypt

REFERENCES:
- [Derived] Abdulrhman MM, El-Hefnawy MH, Aly RH, Shatla RH, Mamdouh RM, Mahmoud DM, Mohamed WS. Metabolic effects of honey in type 1 diabetes mellitus: a randomized crossover pilot study. J Med Food. 2013 Jan;16(1):66-72. doi: 10.1089/jmf.2012.0108. Epub 2012 Dec 20. PMID 23256446
- See also: Faculty of medicine, Ain Shams University, Egypt — http://med.shams.edu.eg/